CLINICAL TRIAL: NCT03817086
Title: Combining Physical and Mental Practice for the Rehabilitation of Upper Extremity Movement Impairments Secondary to Traumatic Brain Injury
Brief Title: Physical and Mental Practice for Bimanual Coordination Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R970-17
Record Dates: First submitted 2019-01-10; First posted 2019-01-25 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Traumatic Brain Injury; Weakness, Muscle; Coordination Impairment
MeSH Terms: conditions — Brain Injuries, Traumatic; Muscle Weakness; Ataxia | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hand coordination and mental practice (Experimental): In a total of 12 training sessions (days), 3 sessions per week over 4 weeks, participants practice physical in-phase and out-of-phase movement of both limbs for 40 minutes. Every 10 minutes, participants get a 2 minutes break during which the participants are asked to mentally imagine doing the task with an action observation of perfect performance.
  Interventions: Behavioral: Hand coordination and mental practice
- Hand coordination and action observation (Active Comparator): In a total of 12 training sessions (days), 3 sessions per week over 4 weeks, participants practice physical in-phase and out-of-phase movement of both limbs for 40 minutes. Every 10 minutes, participants get a 2 minutes break during which the participants are asked to observe a visual feedback of performance.
  Interventions: Behavioral: Hand coordination and action observation

INTERVENTIONS:
Behavioral: Hand coordination and mental practice — 20 chronic (>1year) moderate to severe TBI patients, with upper extremity movement deficits, will be randomly and equally assigned to two groups.
  In the experimental group, participants undergo 5 weeks (3 hrs/week) of physical practice training combined with mental practice (MP group).
  Other Names: experimental group
  Arms: Hand coordination and mental practice
Behavioral: Hand coordination and action observation — In the control group 2, participants undergo 5 weeks (3 hrs/week) of physical training (PP group).
  Other Names: control group
  Arms: Hand coordination and action observation

SUMMARY:
Traumatic Brain Injury (TBI)patients often suffer from loss of muscle strength in the hand and foot, decrease in coordination and high muscle tone (spasticity). In this study, investigators seek to compare how two different training programs can improve the coordination and symptoms of fatigue in individuals with movement deficits secondary to TBI. Using brain imaging, the study will also investigate changes in brain structure and activity associated with hand movement.

DETAILED DESCRIPTION:
Moderate and severe Traumatic Brain Injury (TBI) commonly causes upper extremity physical impairments that persist even after years of injury; these deficits are attributed to damage in brain structure and changes in structural and functional connectivity. Bimanual coordination deficits and muscle weakness have a significant impact on TBI survivors' well-being, and conventional therapy did not provide high success in treating these two issues. The investigators relate this lag in efficiency to two main reasons: 1) absence of outcome measures to quantify these deficits in a clinical setting, and 2) mental and cognitive fatigue and short attention span in TBI survivors, which limits the feasibility to enroll TBI survivors in intensive training protocols.

The investigators long-term goal is to provide effective rehabilitation training to help TBI survivors in regaining proper bimanual coordination of hand movement and higher hand muscles' strength. Mental practice includes motor imagery and action observation, and neural imaging studies have shown that both motor imagery and action observation share similar neural mechanism as movement execution. In addition, interventional studies have shown success in combining physical and mental practice to improve motor function of stroke survivors, and it does not induce muscle fatigue.

Hence, the first aim of this pilot study is to compare the therapeutic efficacy of combining physical practice with mental practice (motor imagery and action observation) (MP) versus physical practice only with action observation (PP) alone to improve hand bimanual coordination and muscle strength of TBI survivors. Twenty subjects will be randomly and equally assigned to either of two training groups. Maximum Voluntary Contraction (MVC), Reaction Time (RT), and Percent of Error in Matching (PEM) a Target will be used as primary outcome measures in addition to functional-based measures (Wolf Motor Function Test WMFT). In addition, activation maps (functional MRI data) will be established for the brain neural networks before and after training. The investigator's second aim is to study if either or both interventions (MP and PP) induce reorganization in brain activity and in functional (at rest) and effective (during a task) connectivity.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 20 to 60 years old.
* have been diagnosed with a moderate to severe Traumatic Brain Injury.
* must have had the injury more than 12 months ago.
* have problems controlling my arm movements.
* right handed.
* speak and understand English.
* willing and able to travel to Kessler Foundation in West Orange, NJ for the 3 testing sessions and the 12 sessions of intervention.
* must have stable health with no expected medication changes for the next 4 months.
* able to understand instructions that are part of the testing and intervention.

Exclusion Criteria:

* have had a penetrating Traumatic Brain Injury.
* have severe spasticity (stiffness and tightness in my muscles) as determined by study staff.
* have had other brain injuries or illnesses in addition to the Traumatic Brain Injury (for example, epilepsy, MS).
* use illegal substances at this time, like drugs
* have had a brain injury that was non-traumatic such as a stroke or brain tumor.
* am enrolled in another research study that is likely to affect my participation in this research study.
* have a history of psychiatric illness (for example, bipolar disorder, schizophrenia, or psychosis).

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Maximum voluntary contraction | Pretest (before training), Posttest (immediately after end of training), Retention test (3 weeks after end of training)
  maximum force exerted by each hand during squeezing a handgrip force sensor
Change in Reaction Time | day 1, day 2, day 3, day 4, day 5, day 6, day 7, day 8, day 9, day 10, day 11, day 12
  Reaction time is the time between real movement, and the time participant was instructed to move. This reaction time will be recorded for every training trial. The average of reaction time in each training day (total 12) will be used to examine the change in performance (slope) across the 12 training days, from day 1 until day 12 of the intervention.
Change in Percent of Error in force matching | day 1, day 2, day 3, day 4, day 5, day 6, day 7, day 8, day 9, day 10, day 11, day 12
  Percent of error is the mismatch between the force exerted by the participant and the required force as per the instructions in each training trial. This Percent of Error will be recorded for every training trial. The average of errors in each training day (total 12) will be used to examine the change (slope) in performance across the 12 sessions (days) of the intervention.
Change in wolf motor function test | Pretest (before training), Posttest (immediately after end of training), Retention test (4 weeks after end of training)
  assessment of upper extremity function
Change in within-brain effective connectivity | Pretest (before training), Posttest (immediately after end of training)
  connectivity between sensorimotor and attention network during inphase and out-phase hand coordination task
Change in resting state function connectivity | Pretest (before training), Posttest (immediately after end of training)
  connectivity between sensorimotor and attention network at rest
Change in brain structural connectivity (DTI) | Pretest (before training), Posttest (immediately after end of training)
  cerebrospinal tract connectivity

SECONDARY OUTCOMES:
stroop effect test | Pretest (before training), Posttest (immediately after end of training), Retention test (3 weeks after end of training)
  neuropsychology assessments of reaction time
trail making test | Pretest (before training), Posttest (immediately after end of training), Retention test (3 weeks after end of training)
  neuropsychology assessments of task switching and visual attention

CONTACTS AND LOCATIONS:
Overall Officials: Soha Saleh, PhD, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No